CLINICAL TRIAL: NCT00537875
Title: Evaluation of the Effect of Zingiber Officinalis on Nausea and Vomiting in Patients Receiving Cisplatin Based Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Institute of Tuberculosis and Lung Disease, Iran (Other Government)
Responsible Party: Principal Investigator, Shadi Baniasadi, associate professor, National Research Institute of Tuberculosis and Lung Disease, Iran
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 5336-18-06-86
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Ginger
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger — Capsule, 1000 mg, BID, 3 days
  Arms: 1
Dietary Supplement: Placebo — Capsule, 1000 mg, BID, 3 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether powdered ginger root (encapsulated ginger) is effective for reducing the frequency, duration and severity of both acute and delayed nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give written informed consent.
* Have a diagnosis of cancer and currently receiving chemotherapy containing cisplatin (any dose).
* Scheduled to receive antiemetics: granisetron (kytril), hydrocortisone.
* Must be able to complete study questionnaires.
* Must be able to swallow capsules.

Exclusion Criteria:

* Have no clinical evidence of current or impending bowel obstruction.
* Concurrent radiotherapy that is classified as high or intermediate risk of causing emesis.
* Pregnant or lactating.
* Patients taking therapeutic doses of coumadin (individuals on low-dose to maintain peripheral or central venous catheters are allowed), aspirin (individuals taking low-dose 80mg aspirin are allowed), or heparin.
* Patients with a history of a bleeding disorder(s) in past 6 months and those experiencing thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Nausea, Vomiting | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Baniasadi, Ph.D., Principal Investigator — National Research Institute of Tuberculosis and Lung Disease (NRITLD)-Shaheed Beheshti University of Medical Sciences
Locations (1):
- National Research Institute of Tuberculosis and Lung Disease (NRITLD), Tehran, Iran